CLINICAL TRIAL: NCT07164014
Title: Dietary Modifications, Like Changing Macronutrient Distribution and Improving Food Quality, Are Main Therapeutic Approaches for Managing Oxidative Stress, Inflammation, and Metabolic Syndrome: Mediterranean Diet is Scientifically Endorsed as Promoting Healthy and Reducing the Risk of Cognitive Decline
Brief Title: The Impact of the Mediterranean Diet on Anthropometric Indices, Lipid Profiles, Energy Metabolism Signaling Proteins and Inflammatory Cytokines in Psychiatric Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ali Abdullah Alyousef, Head Of Clinical Nutrition, King Saud University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 95-EP-2023, KingFahadHospital
Record Dates: First submitted 2025-08-11; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome (MetS); Psychiatric Disorders; Mediterranean Diet; Inflammatory Cytokines; Energy Metabolism; Lipid Profiles
MeSH Terms: conditions — Metabolic Syndrome; Mental Disorders | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The trial included two stages of 8-week intervention periods separated by a 2-week washout period. The hospital kitchen provided the preferred food list, menu, and MD plan design for the patients enrolled in this diet.A certified registered dietician analyzed the data. All 30 psychiatric patients participated in the MD intervention for eight weeks after consuming their regular diets during the washout phase. Following the 14-day washing period, the same group was given a hospitalized diet as a control diet that included medication supplements. An 18-week 2 × 2 crossover design was used in the study. All the anthropometric measurements and blood profiles were performed at baseline (pre-intervention), and after week 8 (post-intervention) after a 10-h overnight fast.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Group 1 (Experimental): The trial is a randomized 2×2 crossover where each participant receives both interventions separated by a washout.
  Interventions:
  Mediterranean Diet - Provided for 8 weeks Hospital Diet - Provided for 8 weeks after a 2-week washout.
  Interventions: Other: Mediterranean diet; Other: Hospital diet
- Arm 2: Group 2 (Experimental): The trial is a randomized 2×2 crossover where each participant receives both interventions separated by a washout.
  Interventions:
  Hospital Diet - Provided for 8 weeks, includes standard hospital meals
  Mediterranean Diet - Provided for 8 weeks after a 2-week washout.
  Interventions: Other: Mediterranean diet; Other: Hospital diet

INTERVENTIONS:
Other: Mediterranean diet — Mediterranean Diet Total Calories: ~1,980 kcal Protein: ~110 g Carbohydrates: ~132 g Fat: ~117 g Diet Type: Mediterranean: Moderate-calorie, high in unsaturated fats, includes fermented dairy Omega-3 Sources: Present: Fish, Olive Oil, Nuts Oil/Fat Types: Olive oil, tahini, nuts (mostly monounsaturated & polyunsaturated)
  Other Names: Arm 1: Group 1; Arm 2: Group 2
Other: Hospital diet — Hospital diet Total Calories: ~3,100 kcal Protein: ~160 g Carbohydrates: ~280 g Fat: ~150 g Diet Type: High Protein, High Calorie: High in saturated fats, refined carbs, and animal proteins Omega-3 Sources: Minimal: Mostly absent Oil/Fat Types: Animal fats (saturated), dairy fat, minimal unsaturated fat
  Other Names: Arm 2: Group 2; Arm 1: Group 1

SUMMARY:
Background: Dietary modifications, like changing macronutrient distribution and improving food quality, are the main therapeutic approaches for managing oxidative stress, inflammation, and metabolic syndrome. Mediterranean diet is scientifically endorsed as promoting healthy aging and reducing the risk of cognitive decline when compared to the Western-style diet pattern. Objective: Analyzing the beneficial effect of the Mediterranean diet (MD) on anthropometric indices, inflammatory markers, lipid profiles in psychiatric patients with metabolic syndrome, compared to the standard hospital diet (HD). Methods: The study was designed as a crossover study; 15 male and 15 female participants with psychiatric disorders were enrolled, and they were intervened with either MD or HD for 8 weeks. Anthropometric parameters, inflammatory cytokines, lipid profile, and metabolic markers were measured with two stages of pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults with psychiatric conditions
* Diagnosed with three components of metabolic syndrome

Exclusion Criteria:

* cognitive or physical impairments that made it difficult to gather all pertinent information
* Non-Hospitalized patients

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Written informed consent was obtained from the participant or their legal guardian on behalf of the study participants.
Enrollment: 144 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Change in Anthropometric measurement | Baseline, Week 8, 11 week, and Week 18
  Four visits were conducted to measure anthropometric parameters using the Tanita Model BC-418® body composition analyzer (Tokyo, Japan). The participants were positioned standing, and electrodes were affixed to their hands and feet. Before the test, participants were allowed to fast for 10 h, and following each measurement, their palms and soles were cleansed. Height (cm), body weight (Kg), body mass index (BMI), abdominal circumference (AC), percentage body fat (PBF), muscle mass percentage (MMP), and visceral fat (VF) were automatically measured by the preprogrammed instrument when it was connected to an ultrasonic height meter.
Blood pressure | Baseline, Week 8, week 11, and Week 18
  Blood pressure was monitored three times a day, specifically between 8:00 am and 10:00 am, 2:00 pm and 4:00 pm, and from 6:00 pm. to 8:00 PM. All hypertensive readings were taken at least 30 minutes following each meal using an Omron HEM-7136 blood pressure monitor (Omron Health Care Co, Ltd, Matsusaka, Japan). Triplicate readings were collected at each time point on the upper right arm with a one-minute interval.
Change in Fasting Blood Glucose | Baseline, Week 8, week 11 and Week 18
  Serum glucose measured via venous blood sample after 10-hour overnight fast, analyzed using automated chemistry analyzer.
Change in Serum Lipid Profile | Baseline, Week 8, week 11 and Week 18
  Total cholesterol, HDL, LDL, and triglycerides measured via enzymatic colorimetric methods.

SECONDARY OUTCOMES:
Changes in Hormones | Baseline, Week 8, week 11 and Week 18
  Insulin, testosterone, serotonin, norepinephrine, thyroid stimulating hormone, thyroxine T4, triiodothyronine T3, prolactin, and cortisol. A standard solution was used to produce a standard curve for all hormones
Change in Inflammatory Markers | Baseline, Week 8, week 11 and Week 18
  Pro-inflammatory cytokines (IL-1β, IL-12, and TNF-α) and anti-inflammatory cytokines (IL-6, IL-10, and IL-31) were quantitatively analyzed using the ELISA method.
  The concentrations of plasma α-melanocyte stimulating hormone (α-MSH), carbohydrate response element binding protein (ChREBP), fibroblast growth factor-21 (FGF-21), and agouti-related protein (AgRP) were also analyzed using the ELISA method following the manufacturer's protocol (Bioassay Technology Laboratory, Shanghai, China).

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No